CLINICAL TRIAL: NCT04192448
Title: The Roles of Acute Alcohol Intoxication, State Anger, and Emotion Regulation on Men's Sexual Aggression Intentions
Brief Title: Men, Mood, and Attention Study: Examination of Alcohol, State Anger, and Emotion Regulation Sexual Aggression
Acronym: MMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Procedures not feasible due to COVID-19 and administrative concerns
Sponsor: Elizabeth C Neilson (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Elizabeth C Neilson, Assistant Professor, Morehead State University
Organization: Morehead State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-10-13; 2P20GM103436 (NIH)
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Intoxication; Anger
Keywords: Sexual Violence; Alcohol consumption
MeSH Terms: conditions — Alcoholic Intoxication; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: The study utilizes a 2x2 (Alcohol and Emotion) design in which participants will be randomly assigned to one of four groups: AlcoholxAnger, AlcoholxControl, SoberxAnger, SoberxControl
Who Masked: Participant
Masking Description: Participant will only be blind to emotion condition. Participants will be informed of their alcohol condition. Investigator and experimenter will be aware of participants' assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AlcoholxAnger (Experimental): Participant will receive alcohol, the dose of which will be administered to result in a BAC of .08%. Participants will also receive an anger emotion induction, in which the experience of frustration and irritability is induced.
  Interventions: Other: Alcohol Administration; Other: Mood Induction
- AlcoholxControl (Experimental): Participant will receive alcohol, the dose of which will be administered to result in a BAC of .08%. Participants will also receive a control emotion induction, in which they are exposed to a neutral mood induction.
  Interventions: Other: Alcohol Administration; Other: Mood Induction
- SoberxAnger (Experimental): Participant will not receive alcohol, therefore their BAC will be .00%. Participants will also receive an anger emotion induction, in which the experience of frustration and irritability is induced.
  Interventions: Other: Alcohol Administration; Other: Mood Induction
- SoberxControl (Sham Comparator): Participant will not receive alcohol, therefore their BAC will be .00%. Participants will also receive a control emotion induction, in which they are exposed to a neutral mood induction.
  Interventions: Other: Alcohol Administration; Other: Mood Induction

INTERVENTIONS:
Other: Alcohol Administration — The clinical trial does not involve any treatment. Participant will be randomly assigned to receive alcohol (BAC = .08%) or water (BAC = .00%).
Other: Mood Induction — The clinical trial does not involve any treatment. Participants will be randomly assigned to receive an anger emotion induction or a control (neutral) mood induction.

SUMMARY:
Given the public health and social relevance of sexual aggression and the gap in the extant literature regarding state anger, emotion regulation, alcohol, and sexual aggression, the present study will contribute to our understanding of emotion regulation's role in sexual aggression perpetration. The proposed 2-year research plan will examine the effects of alcohol intoxication, state anger, and emotion regulation on men's sexual aggression intentions. This study will recruit non-monogamous, men (individuals who identify their gender as male and whose biological sex is male) who have sex with women, ages 21-35. While more research on female perpetrators is needed, the proposed study will exclusively recruit males for the following reasons: 1) the scientific literature indicating the majority of sexually aggressive acts are perpetrated by men; and 2) the current sexual aggression analog has not been piloted with female participants and would require preliminary experiments to determine its appropriateness. The study will utilize a 2x2 design in which participants are randomized to beverage condition [alcohol (target BAC= .08gm%) or control (no alcohol control)] and an emotion induction (anger induction or control). The outcomes will be assessed using a sexual aggression analog which participants will complete on the descending limb of alcohol intoxication and indicate the likelihood that they would engage in various sexually aggressive acts. The study also includes self-report measurements of state anger and emotion regulation to explore emotion regulation as a moderator in the associations among alcohol intoxication, state anger, and sexual aggression intentions.

DETAILED DESCRIPTION:
Males ages 21 to 35 will be recruited from the community through fliers and advertisements in bars and local publications (print and electronic) and instructed to call the lab for telephone screening or complete an online web-screening survey. Sexual aggression is a pervasive and highly prevalent problem on college campuses, so the project will heavily advertise at the local college campus. The screening will include an assessment of typical alcohol consumption patterns, risk for current or past alcohol use disorder, and sexual risk-taking.

Participants (N=180) will be compensated $10 per hour of lab participation for a maximum payment of $80. Participants will begin by completing a series of background measures (see Measures) related to alcohol consumption and expectations, sexual aggression perpetration history, trait anger, and trait emotion regulation. Participants will complete factors of personality that have demonstrated associations with both emotion regulation and sexual aggression as covariates, including psychopathy, sensation seeking, and impulsivity.

Participants will be randomly assigned to receive beverages consisting of either an alcohol dose (target peak BAC =.08gm%) or a control (non-alcoholic) beverage. Participants will be informed into which alcohol condition they have been assigned. Using a double-blind procedure, participants will be block randomized by self-reported sexual aggression perpetration history [(none = no history of perpetration) vs. (low = history of unwanted sexual contact or sexual coercion) vs. (high = attempted or completed perpetration of incapacitated or forced rape)]. A computer algorithm will be used to assign participants to the experimental conditions such that participants with none, low, and high perpetration history are evenly distributed across beverage conditions. Individuals assigned to the alcohol condition will consume a beverage comprised of cranberry juice and 100 proof vodka, while individuals assigned to the control condition will consume a beverage comprised of cranberry juice and water. The total liquid is divided equally between three cups, and participant is given nine minutes to consume the total amount (e.g., three minutes per cup). To ensure stable absorption of alcohol and decrease the likelihood of nausea, the experimenter will instruct the participant to consume the beverages evenly and to avoid drinking quickly. Following beverage administration, participants will be Breathalyzed every five minutes until they attain two Breathalyzer readings of .08%gm to ensure their BAC will descend during the emotion induction and sexual aggression analog. A yoking procedure will be employed for control participants in which each control participant is paired with an alcohol dose participant and receive an equal number of Breathalyzer checks.

Participants will also be randomly assigned to an emotion induction condition consisting of either an anger emotion induction or a control emotion induction. This study will employ deception as individuals will not be told they have been assigned to different emotion induction conditions. The emotion induction consists of two parts: 1) an emotion recall task; and 2) provocation task. Individuals assigned to the anger induction will be instructed to recall an incident in the last 30 days when they felt angry, frustrated, or "pissed off". They will then be given five minutes to write as much as possible about that incident and their response. Participants in the control condition will be instructed to write for five minutes about a neutral topic (e.g., cooking dinner, going for a walk; Marci et al., 2007). The writing samples from all participants will be collected and coded by independent coders to identify whether participants accurately engaged in the task. Following the emotion recall portion of the induction, participants will begin a provocation task. Both groups will begin an attention task. Participants assigned to the anger condition will be given negative feedback about their performance. Participants assigned to the control condition will complete the task without feedback and then will be thanked for their participation.

Upon completion of both portions of the emotion induction, participants will read and project themselves into a written hypothetical sexual situation displayed on a computer. The stimulus story will be approximately 1,600 words and be written at a 5th grade reading level. The story will depict a sexual encounter between the participant and a hypothetical female, in which the female in the story will initially engage in consensual sexual activity however will gradually display and express resistance to engaging in intercourse. Participants will then complete assessment of outcome measures.

Immediately after completing the scenario, participants will be required to watch one of three neutral videos (e.g., comedy clips, nature documentaries) to assist with distancing and detaching from the content of the story. After completing the videos, sober participants will be debriefed and paid for their time. Intoxicated participants will be provided with food, beverages, and entertainment until their BAC descended to below .04%gm. Once their BAC has descended to below .04%gm, these participants will be debriefed and paid for their time.

ELIGIBILITY:
Inclusion Criteria:

* Biologically male and identify their gender as male
* Between the ages of 21-35
* Must be Interested in sexual activity with women
* Must have engaged in at least one instance of sex without a condom in the last six months
* Must on average consume between 5 and 25 standard drinks per week
* Must have previously had an instance of heavy episodic drinking (HED; at least five alcoholic drinks in two hours) in the last six months
* No history of or current alcohol problems (as determined by the Brief Michigan Alcoholism Screening Test)
* No past or current medical condition or take medications which contraindicate alcohol consumption

Exclusion Criteria:

* being in a monogamous relationship of longer than six months or not having sexual intercourse at all within the past six months
* Any history or current alcohol problems (as determined by the Brief Michigan Alcoholism Screening Test)
* Currently taking medications which contraindicate alcohol consumption
* Currently or ever diagnosed with a medical condition that contraindicates alcohol consumption
* Currently enrolled as a student at Morehead State University

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be biologically male participants whose gender identity is male.
Enrollment: 3 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Neilson, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Morehead State University, Morehead, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muehlenhard CL, Peterson ZD, Humphreys TP, Jozkowski KN. Evaluating the One-in-Five Statistic: Women's Risk of Sexual Assault While in College. J Sex Res. 2017 May-Jun;54(4-5):549-576. doi: 10.1080/00224499.2017.1295014. Epub 2017 Apr 4. PMID 28375675
- [Background] Abbey A. Alcohol-related sexual assault: a common problem among college students. J Stud Alcohol Suppl. 2002 Mar;(14):118-28. doi: 10.15288/jsas.2002.s14.118. PMID 12022717
- [Background] Abbey A, Wegner R. Using Experimental Paradigms to Examine Alcohol's Role in Men's Sexual Aggression: Opportunities and Challenges in Proxy Development. Violence Against Women. 2015 Aug;21(8):975-96. doi: 10.1177/1077801215589378. Epub 2015 Jun 5. PMID 26048214
- [Background] DeGue S, Valle LA, Holt MK, Massetti GM, Matjasko JL, Tharp AT. A systematic review of primary prevention strategies for sexual violence perpetration. Aggress Violent Behav. 2014 Jul-Aug;19(4):346-362. doi: 10.1016/j.avb.2014.05.004. PMID 29606897
- [Background] Connor JP, Grier M, Feeney GF, Young RM. The validity of the Brief Michigan Alcohol Screening Test (bMAST) as a problem drinking severity measure. J Stud Alcohol Drugs. 2007 Sep;68(5):771-79. doi: 10.15288/jsad.2007.68.771. PMID 17690811
- [Background] Martin CS, Sayette MA. Experimental design in alcohol administration research: limitations and alternatives in the manipulation of dosage-set. J Stud Alcohol. 1993 Nov;54(6):750-61. doi: 10.15288/jsa.1993.54.750. PMID 8271813
- [Background] Giancola PR, Zeichner A. The biphasic effects of alcohol on human physical aggression. J Abnorm Psychol. 1997 Nov;106(4):598-607. doi: 10.1037//0021-843x.106.4.598. PMID 9358690
- [Background] Davis KC, George WH, Norris J, Schacht RL, Stoner SA, Hendershot CS, Kajumulo KF. Effects of alcohol and blood alcohol concentration limb on sexual risk-taking intentions. J Stud Alcohol Drugs. 2009 Jul;70(4):499-507. doi: 10.15288/jsad.2009.70.499. PMID 19515289
- [Background] Laber EB, Shedden K. Statistical Significance and the Dichotomization of Evidence: The Relevance of the ASA Statement on Statistical Significance and p-values for Statisticians. J Am Stat Assoc. 2017;112(519):902-904. doi: 10.1080/01621459.2017.1311265. Epub 2017 Oct 30. No abstract available. PMID 29348701
- See also: Recommended council guidelines on ethyl alcohol administration in human experimentation — http://www.niaaa.nih.gov/research/guidelines-and-resources/administering-alcohol-human-studies

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study began in September 2020 after IRB approval was obtained for study modifications necessary to comply with COVID-related safety precautions. Advertisements were placed in local business, emphasizing alcohol-serving establishments, and authorized posting areas in local community colleges and four-year universities. Online advertisements were posted in social media sites (e.g., Facebook, Instagram) and forums (e.g., Reddit, Craiglist). Recruitment continued until May 2021.
Pre-assignment Details: After enrollment, participants completed baseline measures. Participants were block randomized to condition arm based upon their past sexual assault perpetration status, such that an equal number of participants who had previously perpetrated sexual assault were assigned to each condition arm. No participants were excluded prior to group assignment.
Period: Overall Study
Arm/Group | AlcoholxAnger | AlcoholxControl | SoberxAnger | SoberxControl
Started | 1 | 1 | 0 | 1
Completed | 1 | 1 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population met all the inclusion criteria as outlined in the initial proposal, thus were cisgender men who engaged in moderate to heavy drinking and sexual risk-taking. The number enrolled is substantively different than proposed due to administrative barriers to the study and COVID-related barriers that impacted recruitment (closure of alcohol-serving establishments, community concern regarding participation in in-person studies during the pandemic).
Groups:
- Total: Total of all reporting groups
Arm/Group | AlcoholxAnger | AlcoholxControl | SoberxAnger | SoberxControl | Total
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (0) | 35 (0) |  | 30 (0) | 32 (2.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 0 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants selected the race with which they identified: Native American or American Indian, Asian or South Asian, Black or African American, Native Hawaiian or Pacific Islander, White, Multiracial or Biracial, Latino/Hispanic, and Not Listed (with an option to write in a race). While Latino/Hispanic category is most typically conceptualized as an ethnicity, not a racial identity, this category was required by the IRB. Participants could choose more than one category and if so, were classified as Multiracial. A separate question asked if participants identified as Latino/Hispanic (Yes/No).
  Participants
    Race and Ethnicity: White/Non-Latino | 1 | 1 | 0 | 0 | 2
    Race and Ethnicity: Black or African American/Non-Latino | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — All data collection occurred in the United States
  Participants
    United States | 1 | 1 | 0 | 1 | 3
Sexual Experiences Survey [Mean (Standard Deviation); unit: units on a scale] — The SES assesses a range of sexually aggressive acts and tactics perpetrated against another person who has not consented to those acts. Participants indicated the number of times that a tactic or multiple tactics were used up to 3 times. Scores are computed such that a participant's score reflects the most severe sexually aggressively act they have perpetrated since age 14 (0 = None; 1 = unwanted sexual contact by any tactic; 2 = Attempted rape by coercion; 3 = Rape by coercion; 4 = Attempted rape by incapacitation or force; 5 = Rape by incapacitation or force)
  units on a scale | 3 (0) | 0 (0) |  | 4 (0) | 2.33 (2.08)
Difficulties in Emotion Regulation Scale [Mean (Standard Deviation); unit: units on a scale] — The Difficulties in Emotion Regulation Scale is a 36-item, self report of problems with emotional acceptance, emotional awareness, emotional clarity, access to emotion regulation strategies, difficulties with impulse control, and difficulties engaging in goal directed behavior when experience intense emotions. Scores range from 36 to 180. Higher scores indicate greater difficulties with emotion regulation. Individuals scoring above 108 indicate difficulties regulating their emotions more than half of the time.
  units on a scale | 88 (0) | 62 (0) |  | 73 (0) | 74.33 (13.05)

OUTCOME MEASURES:

1. Primary Outcome: Sexual Aggression Intentions
Description: Mean score of 22 items assessing behavioral intentions (1 = Not at Likely to 7 = Very Likely) to act sexually aggressively against a hypothetical female
Time Frame: 20 minutes
Population: The population analyzed is comprised of the three participants who were enrolled into the study. No participants were analyzed in the Sober x Anger arm because no participants were randomly assigned to that arm.
Measure: Number; unit: score on a scale
Arm/Group | AlcoholxAnger | AlcoholxControl | SoberxAnger | SoberxControl
Number analyzed (Participants) | 1 | 1 | 0 | 1
score on a scale | 2.18 | 4.73 |  | 1.64
Statistical Analysis 1: Comparison: AlcoholxAnger vs AlcoholxControl vs SoberxControl; The number of participants enrolled in the study constrained the type of statistical analyses able to be conducted. Indeed, the Sober x Anger condition could not be compared to the other arms because no participants were randomly assigned to that arm; Test type: Other — Target sample size was 200 participants. Power calculation was determined using nQuery version 8.4.1 for the 2x2 design, using 50 subject per group (including a conservative 10% dropout). Power calculation estimated 80% power to detect an effect size of 0.3 in both factors with no interaction, and greater power if there is an interaction effect. Current enrollment indicates study is underpowered. Because there are not enough participants to conduct an ANOVA or ANCOVA, t-tests were conducted; p = .28, t-test, 1 sided; This t-test examined the difference in sexual aggression intentions between those in the Alcohol condition and those in the Sober condition; Mean Difference (Final Values) = 1.82, 95% CI 2-sided [-29.82 to 26.19] — The estimation parameter refers to the mean difference in the outcome between those in the Alcohol condition and those in the Sober condition. A positive value indicates greater likelihood of sexual aggression among those in the Alcohol condition
Statistical Analysis 2: Comparison: AlcoholxAnger vs AlcoholxControl vs SoberxControl; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .39, t-test, 1 sided; This t-test examined the difference in sexual aggression intentions between those in the Anger condition and those in the Control condition; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-33.01 to 35.01] — The estimation parameter refers to the mean difference in the outcome between those in the Anger condition and those in the Control condition. A negative value indicates greater likelihood of sexual aggression among those in the Control condition

2. Secondary Outcome: Physical Aggression Intentions
Description: Mean score of 5 items assessing behavioral intentions (1 = Not at All to 7 = Extremely) of intentions to act physically aggressively against a hypothetical female
Time Frame: 20 minutes
Population: The population analyze dis comprised of the three participants who were enrolled into the study. No participants were analyzed in the Sober x Anger arm because no participants were randomly assigned to that arm.
Measure: Number; unit: score on a scale
Arm/Group | AlcoholxAnger | AlcoholxControl | SoberxAnger | SoberxControl
Number analyzed (Participants) | 1 | 1 | 0 | 1
score on a scale | 1.0 | 1.25 |  | 1.0
Statistical Analysis 1: Comparison: AlcoholxAnger vs AlcoholxControl vs SoberxControl; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .33, t-test, 1 sided; This t-test examined the difference in physical aggression intentions between those in the Alcohol Condition and those in the Sober condition; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-2.88 to 2.63] — The estimation parameter refers to the mean difference in the outcome between those in the Alcohol condition and those in the Sober condition. A positive value indicates greater likelihood of physical aggression among those in the Alcohol condition
Statistical Analysis 2: Comparison: AlcoholxAnger vs AlcoholxControl vs SoberxControl; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .33, t-test, 1 sided; The t-test examined the difference in physical aggression intentions between those in the Anger condition and those in the Control condition; Mean Difference (Final Values) = -.25, 95% CI 2-sided [-2.53 to 2.88] — The estimation parameter refers to the mean difference in the outcome between those in the Anger condition and those in the Control condition. A negative value indicates greater likelihood of physical aggression among those in the Control condition

3. Secondary Outcome: Psychological Aggression Intentions
Description: Mean score of 3 items assessing behavioral intentions (1 = Not at All to 7 = Extremely) of intentions to act psychologically aggressively against a hypothetical female
Time Frame: 20 minutes
Population: The population analyzed is compromised of the three participants who were enrolled into the study. No participants were analyzed in the Sober x Anger arm because no participants were randomly assigned to that arm.
Measure: Number; unit: score on a scale
Arm/Group | AlcoholxAnger | AlcoholxControl | SoberxAnger | SoberxControl
Number analyzed (Participants) | 1 | 1 | 0 | 1
score on a scale | 1.67 | 2.33 |  | 1.33
Statistical Analysis 1: Comparison: AlcoholxAnger vs AlcoholxControl vs SoberxControl; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .23, t-test, 1 sided; The t-test examined differences in psychological aggression intentions between those in the Alcohol condition and those in the Sober condition; Mean Difference (Final Values) = .67, 95% CI 2-sided [-8.00 to 6.67] — The estimation parameter refers to the mean difference in the outcome between those in the Alcohol condition and those in the Sober condition. A positive value indicates greater likelihood of psych aggression among those in the Alcohol condition
Statistical Analysis 2: Comparison: AlcoholxAnger vs AlcoholxControl vs SoberxControl; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .44, t-test, 1 sided; The t-test examined the difference in psychological aggression intentions between those in the Anger condition and those in the Control condition; Mean Difference (Final Values) = -.17, 95% CI 2-sided [-10.84 to 11.17] — The estimation parameter refers to the mean difference in the outcome between those in the Alcohol condition and those in the Sober condition. A negative value indicates greater likelihood of psych aggression among those in the Control condition

ADVERSE EVENTS:
Time Frame: Adverse event data were directly collected during the course of a participant's engagement in the study, which was approximately 5 to 7 1/2 hours. Participants were provided with contact information for the research team and IRB and encouraged to contact either the PI or IRB if they believed they had been negatively affected by the study. The PI monitored study email and voicemail for 1 year.
Description: An adverse event was defined as any unfavorable medical occurrence in a participant temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. A serious adverse event would be one that required immediate medical attention at a hospital emergency room and/or a persistent or significant disruption to functioning or requiring services that would prevent a serious adverse event.
Arm/Group | AlcoholxAnger | AlcoholxControl | SoberxAnger | SoberxControl
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The most notable limitation to the current study is the sample size. The study was terminated after three participants were enrolled from October 2020 to May 2021. Extensive efforts were undertaken to improve recruitment, however administrative limitations placed upon the study by the institution and the ongoing COVID-19 pandemic presented barriers to recruitment. While the Results presented indicate the scores obtained from the data, the sample is too small to draw any meaningful conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT04192448/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04192448/ICF_001.pdf